CLINICAL TRIAL: NCT07267507
Title: Accessory Movements and Associated Factors During Active Cervical Range of Motion
Status: Active, not recruiting | Type: Observational
Sponsor: Atılım University (Other)
Responsible Party: Principal Investigator, Nagihan Acet, Asst. Prof., Atılım University
Other Study IDs: Atılım University-25
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Asymptomatic Condition; Neck Pain
Keywords: Cervical Vertebrae; Range of Motion; Pain; Sleep; Depression
MeSH Terms: conditions — Asymptomatic Diseases; Neck Pain; Pain; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Proprioceptive Dysfunction Group: Individuals with proprioceptive error (more than 4 degree)
- Non-Error Group: Individuals without proprioceptive error-less than 4 degree

SUMMARY:
This project aims to quantify accessory movements that occur during cervical range of motion (ROM) assessment in young adults and to examine their relationship with functional and psychological factors. Although cervical ROM is widely used in clinical practice, accurate measurement is challenged by the complex anatomy of the cervical spine and coupled movements, which may alter true motion values. Despite their clinical relevance, accessory movements have been largely overlooked in both research and routine assessment.

This cross-sectional observational study will include volunteers aged 18-30 years, recruited between January and August 2025 following ethical approval. Individuals with cervical trauma or surgery, neurological disease, recent treatment, musculoskeletal injury, or medications affecting movement will be excluded. Accessory movements will be measured using the CROM device while participants perform flexion-extension, lateral flexion, and rotation, maintaining end-range for 20 seconds to record primary and accessory motions.

Clinical outcomes will include cervical disability (Neck Disability Index), pain intensity (Visual Analog Scale), cervical mechanosensitivity (pressure algometry at the upper trapezius and C2-C7 regions), psychological status (Depression, Anxiety, Stress Scale-21), and sleep quality (Pittsburgh Sleep Quality Index).

DETAILED DESCRIPTION:
Range of motion (ROM) is a routinely accepted parameter used by physiotherapists and other health professionals in the evaluation of spinal movements, serving as both a baseline and outcome measure for documenting disability and the effects of interventions, as well as for adjusting physiotherapy treatment plans. However, due to the complex anatomy of the cervical spine and its associated movements, accurate measurement of cervical ROM remains challenging.

A variety of tools have been developed to assess cervical mobility, ranging from simple visual inspection to advanced three-dimensional motion analysis systems, including goniometers, inclinometers, CROM devices, Optotrak and Vicon systems, radiographic techniques, and smartphone applications.

The anatomy of the cervical spine and the presence of "coupled movements" make the measurement of cervical ROM particularly difficult. Coupled movements refer to accessory motions that accompany a primary target movement. For example, when an individual flexes the head forward while simultaneously rotating it laterally, flexion is considered the primary movement, whereas the accompanying lateral flexion and axial rotation are accessory movements. The complex structure of the functional units of the cervical spine permits the combination of multi-axial movements rather than isolated single-axis motions. Movements of adjacent vertebrae are guided by the geometry of the articular surfaces, which allows the combination of ipsilateral rotation with lateral flexion. At the lower cervical levels, the orientation of the apophyseal joints and the presence of cervical lordosis may lead lateral flexion to be accompanied by ipsilateral rotation and slight extension. Other studies have emphasized the variability in movement patterns that arise due to the presence of these coupled motions, even during simple tasks. Additionally, research has demonstrated that accessory movements can cause substantial variation in the magnitude of the primary movement.

At the structural level of the cervical spine, multiple movement strategies may be used to achieve a specific functional goal. The number of studies describing accessory movements as involuntary patterns developed in the presence of cervical pain is limited, and those that exist vary depending on the measurement technique and participant characteristics. By revealing the impact of often-neglected accessory movements during the assessment of active cervical ROM, the present project aims to introduce conceptual and methodological innovations to cervical mobility evaluation methods. Considering the scarcity of research on this topic, the proposed project will provide a unique contribution to clinical assessment and treatment strategies.

To the best of our knowledge, although there are a limited number of studies investigating the presence of accessory movements during cervical ROM measurement, no research has explored the factors associated with these movements. A better understanding of the characteristics of ROM impairments may help clarify the clinical significance of these relationships. However, in both the literature and clinical practice, the magnitude of accessory movements occurring during cervical ROM has generally been overlooked. The present project addresses this important gap by quantifying accessory movements and, for the first time, comprehensively examining their relationship with both physical and psychological limitations in young individuals. In this context, the project is expected to contribute to the development of more specific and individualized treatment algorithms for individuals with cervical spine dysfunction.

ELIGIBILITY:
Inclusion Criteria:Participants will be included if they:

Are between 18 and 30 years of age

Volunteer to participate in the study

Provide written informed consent.

Exclusion Criteria:Participants will be excluded if they have:

A history of cervical trauma

A history of cervical spine surgery

Any neurological disorder

Received treatment related to the cervical region within the past 6 months

Any musculoskeletal injury that may affect cervical movement

Use of medications that could influence movement or neuromuscular function.

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of young adults aged 18-30 years who volunteer to participate and meet the inclusion criteria. Only individuals without cervical trauma, surgery, neurological disorders, recent treatment, musculoskeletal injuries, or medication use affecting cervical movement will be included, ensuring a homogeneous non-clinical sample suitable for accurately evaluating accessory cervical movements.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Assessment of Accessory Movements | 0-18 months
  Accessory movements occurring during active cervical ROM will be evaluated using the Cervical Range of Motion (CROM) device. In a seated position, the participant's neutral resting posture will first be recorded. Subsequently, they will be instructed to perform flexion, extension, right lateral flexion, left lateral flexion, right rotation, and left rotation in sequence. At the end of each movement, participants will hold the end position for 20 seconds, during which the primary movement and the accessory movements occurring in the other two planes will be recorded.
Assessment of Cervical Disability | 0-18 months
  Cervical disability will be assessed using the Neck Disability Index (NDI), a widely used instrument for evaluating cervical spine dysfunction. The NDI consists of 10 items that measure the impact of neck-related problems on daily activities, including pain intensity, personal care, lifting, reading, headaches, concentration, work status, driving, sleep, and recreational activities. Each item is scored on a scale from 0 to 5, resulting in a total score ranging from 0 to 50. A score of 0 indicates no disability or functional limitation, whereas a score of 50 reflects severe functional impairment. It is recommended that the total score be converted into a percentage, interpreted as follows: 0-4 (no disability), 5-14 (mild disability), 15-24 (moderate disability), 25-34 (severe disability), and 35-50 (complete or very severe disability).
Assessment of Pain Intensity | 0-18 months
  Pain intensity will be assessed using the Visual Analog Scale (VAS). The VAS consists of a 10-cm (100-mm) horizontal line anchored by the descriptors "no pain" at one end and "worst imaginable pain" at the other. Participants will mark the point on the line that represents the intensity of pain they experience, and the distance in millimeters from the "no pain" anchor to the marked point will be recorded as the pain score.
Assessment of Cervical Mechanosensitivity | 0-18 months
  Cervical muscle mechanosensitivity will be evaluated using a pressure algometer (Baseline Force Gauge Model 12-0304; Baseline, NY, USA). The device applies force perpendicular to the tissue through a 0.5 cm² probe at an approximate rate of 3 N/s. With the participant seated, pressure will be applied bilaterally to the midpoint of the upper trapezius muscle and to points located 2 cm lateral to the C2 and C7 articular pillars. Pressure algometry has demonstrated high intra-rater (ICC = 0.94-0.97) and inter-rater reliability (ICC = 0.79-0.90) in individuals with neck pain.
  Participants will be instructed to indicate the moment when the pressure sensation first becomes uncomfortable. This value, defined as the pressure pain threshold (PPT), will be recorded twice with at least 30 seconds between trials, and the mean of the two measurements will be used for analysis.
Assessment of Depression, Anxiety, and Stress: | 0-18 months
  Depression, anxiety, and stress levels will be assessed using the Depression, Anxiety, and Stress Scale-21 (DASS-21). The DASS-21 consists of three subscales-depression, anxiety, and stress-each comprising 7 items. Scores for each subscale are summed and then multiplied by two, yielding a maximum possible score of 42 per domain. Higher scores indicate greater symptom severity. Recommended cut-off ranges vary for each construct: for depression, 0-9 (normal) to ≥28 (extremely severe); for anxiety, 0-7 (normal) to ≥20 (extremely severe); and for stress, 0-14 (normal) to ≥34 (extremely severe).
Assessment of Sleep Disturbances | 0-18 months
  Sleep disturbances will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 19-item questionnaire designed to evaluate sleep habits over the past month and comprises seven components. The total score ranges from 0 to 21, with higher scores indicating poorer sleep quality. A global score of 5 or above is considered indicative of sleep disturbance.

CONTACTS AND LOCATIONS:
Locations (1):
- Atılım University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ağargün, M.Y., H. Kara, and Ö. Anlar, The validity and reliability of the Pittsburgh Sleep Quality Index. Turk Psikiyatri Derg, 1996. 7(2): p. 107-15.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Sariçam, H., The psychometric properties of Turkish version of Depression Anxiety Stress Scale-21 (DASS-21) in health control and clinical samples. Journal of Cognitive Behavioral Psychotherapies and Research, 2018. 7(1): p. 19.
- [Background] Lovibond, S.H., Manual for the depression anxiety stress scales. Sydney psychology foundation, 1995.
- [Background] McCormack HM, Horne DJ, Sheather S. Clinical applications of visual analogue scales: a critical review. Psychol Med. 1988 Nov;18(4):1007-19. doi: 10.1017/s0033291700009934. PMID 3078045
- [Background] Vernon H, Mior S. The Neck Disability Index: a study of reliability and validity. J Manipulative Physiol Ther. 1991 Sep;14(7):409-15. PMID 1834753
- [Background] Aslan E, Karaduman A, Yakut Y, Aras B, Simsek IE, Yagly N. The cultural adaptation, reliability and validity of neck disability index in patients with neck pain: a Turkish version study. Spine (Phila Pa 1976). 2008 May 15;33(11):E362-5. doi: 10.1097/BRS.0b013e31817144e1. PMID 18469684
- [Background] Law EY, Chiu TT. Measurement of cervical range of motion (CROM) by electronic CROM goniometer: a test of reliability and validity. J Back Musculoskelet Rehabil. 2013;26(2):141-8. doi: 10.3233/BMR-2012-00358. PMID 23640315
- [Background] Lysell E. Motion in the cervical spine. An experimental study on autopsy specimens. Acta Orthop Scand. 1969:Suppl 123:1+. doi: 10.3109/ort.1969.40.suppl-123.01. No abstract available. PMID 4907116
- [Background] Harrison DE, Harrison DD, Cailliet R, Janik TJ, Troyanovich SJ. Cervical coupling during lateral head translations creates an S-configuration. Clin Biomech (Bristol). 2000 Jul;15(6):436-40. doi: 10.1016/s0268-0033(99)00098-4. PMID 10771122
- [Background] Boussion, L. and L. Chèze, Étude cinématique tridimensionnelle du rachis cervical: Comparaison entre sujets asymptomatiques et "pathologiques". Kinésithérapie, la Revue, 2011. 11(109-110): p. 36-37.
- [Background] Mangone M, Bernetti A, Germanotta M, Di Sipio E, Razzano C, Ioppolo F, Santilli V, Venditto T, Paoloni M. Reliability of the Cervical Spine Device for the Assessment of Cervical Spine Range of Motion in Asymptomatic Participants. J Manipulative Physiol Ther. 2018 May;41(4):342-349. doi: 10.1016/j.jmpt.2018.01.003. PMID 29751851
- [Background] Cuesta-Vargas AI, Galan-Mercant A, Williams JM. The use of inertial sensors system for human motion analysis. Phys Ther Rev. 2010 Dec;15(6):462-473. doi: 10.1179/1743288X11Y.0000000006. PMID 23565045
- [Background] Tucci SM, Hicks JE, Gross EG, Campbell W, Danoff J. Cervical motion assessment: a new, simple and accurate method. Arch Phys Med Rehabil. 1986 Apr;67(4):225-30. PMID 3964055
- [Background] Frost M, Stuckey S, Smalley LA, Dorman G. Reliability of measuring trunk motions in centimeters. Phys Ther. 1982 Oct;62(10):1431-7. doi: 10.1093/ptj/62.10.1431. PMID 7122701
- [Background] Sukari AAA, Singh S, Bohari MH, Idris Z, Ghani ARI, Abdullah JM. Examining the Range of Motion of the Cervical Spine: Utilising Different Bedside Instruments. Malays J Med Sci. 2021 Apr;28(2):100-105. doi: 10.21315/mjms2021.28.2.9. Epub 2021 Apr 21. PMID 33958964
- [Background] Audette I, Dumas JP, Cote JN, De Serres SJ. Validity and between-day reliability of the cervical range of motion (CROM) device. J Orthop Sports Phys Ther. 2010 May;40(5):318-23. doi: 10.2519/jospt.2010.3180. PMID 20436238
- [Background] Yoon TL, Kim HN, Min JH. Validity and Reliability of an Inertial Measurement Unit-based 3-Dimensional Angular Measurement of Cervical Range of Motion. J Manipulative Physiol Ther. 2019 Jan;42(1):75-81. doi: 10.1016/j.jmpt.2018.06.001. PMID 31054596
- [Background] Jonas R, Demmelmaier R, Hacker SP, Wilke HJ. Comparison of three-dimensional helical axes of the cervical spine between in vitro and in vivo testing. Spine J. 2018 Mar;18(3):515-524. doi: 10.1016/j.spinee.2017.10.065. Epub 2017 Oct 23. PMID 29074465
- [Background] de Koning CH, van den Heuvel SP, Staal JB, Smits-Engelsman BC, Hendriks EJ. Clinimetric evaluation of active range of motion measures in patients with non-specific neck pain: a systematic review. Eur Spine J. 2008 Jul;17(7):905-21. doi: 10.1007/s00586-008-0656-3. Epub 2008 Apr 22. PMID 18427843